CLINICAL TRIAL: NCT03155334
Title: Understanding Evaluation of Patient Information Sheets of Two Multiple Sclerosis Studies Through User Testing Method in a Randomized, Open Label, Crossover Design
Brief Title: Understanding Evaluation of Patient Information Sheets by User Testing Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FISM 2012R2
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: MS (Multiple Sclerosis)
Keywords: Multiple Sclerosis; Patient Information Sheet; User Testing
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevalence of CCSVI in MS (Other): Subjects with prevalence of CCSVI in Multiple Sclerosis and in Other Neurodegenerative Diseases - PIS User Testing
  Interventions: Other: PIS User Testing
- BVD Exploited Against MS (Other): Subjects suffering from Brain venous drainage exploited against Multiple Sclerosis - PIS User Testing
  Interventions: Other: PIS User Testing

INTERVENTIONS:
Other: PIS User Testing — PIS User Testing based on an iterative 4-step process in a cohort of participants (the target group):
  * individual reading of the text;
  * individual questionnaire for a quantitative and qualitative evaluation;
  * a brief semi-structured interview to each participant;
  * a text revision to address any problems identified from participant feedback.

SUMMARY:
The purpose of this randomized, open label, crossover, single site study is to compare the PISs of two Multiple Sclerosis clinical trials to elucidate potential aspects of the given written information that could impact on the smooth running of the studies.

DETAILED DESCRIPTION:
The participation to a clinical trial is based on two forms of information: the spoken information, usually given by a clinician during the enrolment meeting, and the written information, reported on the Participant Information Sheet (PIS). Numerous studies performed to improve and enhance informed consent, have used different methods to evaluate the quality of the given information such as: interview, checklist, questionnaire, readability formulae. Even if these tools can be useful, they show evident limits in detecting the real efficacy of the proposed consent form in terms of the patient's comprehension.

User Testing (UT) is a method originally developed in the 1990 in Australia, to assess how a text about medicinal products performs with its intended users and not just its content.

Generally, the UT is based on an iterative 4-step process in a cohort of participants (the target group):

* individual reading of the text;
* individual questionnaire for a quantitative and qualitative evaluation;
* a brief semi-structured interview to each participant;
* a text revision to address any problems identified from participant feedback; Then the revised document is tested again with a second cohort and this iterative process continues until all issues with the document are resolved. However, a methodological issue not yet explored is whether the UT could be used to compare two different PISs, in order to elucidate aspects that could be involved in improving or worsening the understanding of a PIS.

UT has been recently used to evaluate the PIS belonging to phase I and phase III clinical trials (CT) in Myeloid Leukemia, immunomodulatory therapy and for poor responders in vitro fertilization. To date, in no case the UT method has been tested in patients affected by chronic disease like Multiple Sclerosis (MS).

We want to apply the UT approach to highlight the critical issues and communication difficulties present in PISs used in MS clinical trials.

ELIGIBILITY:
Inclusion Criteria: PwMS (60%) and Caregivers (40%):

for PwMS:

* 18 years or older;
* MS diagnosis according to McDonald criteria;
* Informed consent to the present study for caregivers:
* 18 years or older;
* in being a person who takes care of a PwMS;
* Informed consent to the present study

Exclusion Criteria:

- not having taken part in one of the following trials evaluated in the present study: A) Observational Study of the Prevalence of CCSVI in Multiple Sclerosis and in Other Neurodegenerative Diseases (PIS-A); B) BRAin VEnous DRainage Exploited Against Multiple Sclerosis (PIS-B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
percentage of found and understood-if-found items | 1 day
  percentage

SECONDARY OUTCOMES:
understanding of the text expressed by subject | 1 day
  Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Alberto Battaglia, Prof., Study Director — Fondazione Italiana Sclerosi Multipla (FISM), Genova , (Italy)
Locations (2):
- Fondazione Italiana Sclerosi Multipla (FISM), Genoa, Liguria, Italy
- Opera Contract Research Organization SRL, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Raynor DK. User testing in developing patient medication information in Europe. Res Social Adm Pharm. 2013 Sep-Oct;9(5):640-5. doi: 10.1016/j.sapharm.2013.02.007. Epub 2013 Apr 10. PMID 23583081
- [Background] Knapp P, Raynor DK, Silcock J, Parkinson B. Performance-based readability testing of participant materials for a phase I trial: TGN1412. J Med Ethics. 2009 Sep;35(9):573-8. doi: 10.1136/jme.2008.026708. PMID 19717698
- [Background] Knapp P, Raynor DK, Silcock J, Parkinson B. Performance-based readability testing of participant information for a Phase 3 IVF trial. Trials. 2009 Sep 1;10:79. doi: 10.1186/1745-6215-10-79. PMID 19723335
- [Background] Knapp P, Raynor DK, Silcock J, Parkinson B. Can user testing of a clinical trial patient information sheet make it fit-for-purpose?--a randomized controlled trial. BMC Med. 2011 Jul 21;9:89. doi: 10.1186/1741-7015-9-89. PMID 21777435
- See also: Observational Study of the Prevalence of CCSVI in Multiple Sclerosis and in Other Neurodegenerative Diseases (COSMO), ClinicalTrials.gov Identifier: NCT01384825 — http://clinicaltrials.gov/ct2/show/NCT01384825?term=Cosmo&rank=8
- See also: BRAin VEnous DRainage Exploited Against Multiple Sclerosis (BRAVE-DREAMS), ClinicalTrials.gov Identifier: NCT01371760 — http://clinicaltrials.gov/ct2/show/NCT01371760?term=BRAVE-DREAMS&rank=1